CLINICAL TRIAL: NCT07387328
Title: Validation of New sEMG Electrode Placement Guidelines for the Triceps Surae in Post-stroke Individuals.
Acronym: Vest-P
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Vrije Universiteit Brussel (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2025-0433; 11PKX24N (Other Grant/Funding Number: Research foundation Flanders)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Surface electromyography; guidelines; SENIAM; 3D freehand ultrasound
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons after stroke.

SUMMARY:
Background and rationale:

Surface electromyography (EMG) is a non-invasive method to measure muscle activity, among others in people after a stroke during gait analysis. Measurement quality is strongly influenced by electrode placement. However, the commonly used SENIAM guidelines do not take individual variations in muscle morphology into account, which can lead to inaccurate measurements. In previous research (De Vlieger et al. 2025, Journal of Electromyography and Kinesiology), we demonstrated that the standard placement on the triceps surae (medial and lateral gastrocnemius and soleus) was suboptimal at the group level and sometimes even problematic at the individual level. Therefore, we developed new placement guidelines (EPICA guidelines, Electrode Placement for Individual Calf Anatomy), which are currently being tested in healthy individuals.

Method:

In this project, we aim to validate these guidelines in people after a stroke who exhibit atrophy of their calf muscles. For each participant, electrode positions on the hemiplegic side will be determined according to our guidelines while the participant is lying prone. We will use circular stickers instead of actual EMG electrodes. Stickers will be placed according to the EPICA guidelines (researcher Daan De Vlieger) as well as according to SENIAM. Subsequently, the muscle borders of the triceps surae will be identified on the participant's leg using 2D ultrasound. We will measure the distance between the electrodes and the surrounding muscle borders to map electrode placement on the muscle and thus validate the guidelines.

In the second part of this study, 3D ultrasound recordings will be made of the soleus, medial gastrocnemius, and lateral gastrocnemius with the electrodes (stickers) on these muscles, so that during image processing, electrode positions can be visualized relative to the entire muscle, including in depth. In addition, participants who can safely walk without an ankle-foot orthosis will be asked to walk a maximum of five times ten meters. Additionally, an ultrasound probe will be attached to the leg to investigate how the electrode position relates to the muscle-tendon junction during movement. Subsequently, actual electrodes will also be placed to record muscle activity during walking and heel raises.

Furthermore, all participants will be asked to do a heel raise to activate the calf muscles. In this way, we will evaluate whether our guidelines also lead to optimal placement for reliable and high-quality EMG signals in this patient group. We will also administer the Fugl-Meyer Assessment of the lower limb, measure passive ankle range of motion with a goniometer, and measure lower leg length with a tape measure. These will be used as descriptive parameters of our study population.

Patients will be asked on a voluntary basis to participate in a second, short measurement approximately two weeks after the first session. During this measurement, electrode placement will again be performed according to the EPICA guidelines. 2D ultrasound will again be used to calculate the distances between the electrodes and the muscle borders. This second measurement is necessary to investigate the test-retest reliability of the EPICA guidelines in people after a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals who have experienced a stroke (CVA or cerebrovascular accident).
* Have no other neurological disorder.
* Are able to lie in the prone position for approximately one and a half hours.
* Are able to walk without shoes for the walking component (only applicable to participants who will perform walking). The use of an assistive device such as a walking stick (or similar) is permitted.

Exclusion Criteria:

* Presence of other neurological or orthopedic conditions that may influence the measurements and results (e.g., Parkinson's disease, peripheral neuropathy of the lower limbs, severe ankle osteoarthritis limiting range of motion, etc.).
* Having undergone a surgical intervention on the hemiparetic lower leg (e.g., ankle joint arthrodesis, etc.).
* Severe cognitive impairments that prevent understanding participation in the study (assessed using the AbilityQ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons after stroke.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Electrode-muscle boundary distances for EPICA-electrodes | At study enrollment and a second time at least two weeks later.
  These distances, measured with a tape measure, will be obtained between the EPICA electrode positions and the muscle boundaries as visualized using 2D ultrasound.
Electrode-muscle boundary distances for SENIAM-electrodes | At study enrollment.
  These distances, measured with a tape measure, will be obtained between the SENIAM electrode positions and the muscle boundaries as visualized using 2D ultrasound.
Triceps surae muscle geometry | At study enrollment.
  Triceps surae muscle geometry will be measured using 3D freehand ultrasound.
Muscle-tendon junction displacement of the lateral gastrocnemius during walking. | At study enrollment.
  This will be measured with dynamic 2D ultrasound.
Muscle-tendon junction displacement of the lateral gastrocnemius during a heel raise. | At study enrollment.
  This will be measured using dynamic 2D ultrasound.
Muscle-tendon junction displacement of the medial gastrocnemius during walking. | At study enrollment.
  This will be measured using dynamic 2D ultrasound.
Muscle-tendon junction displacement of the medial gastrocnemius during a heel raise. | At study enrollment.
  This will be measured using dynamic 2D ultrasound.
Quality features of the surface electromyography signals obtained from the EPICA electrodes during the dynamic tasks. | At study enrollment.
Quality features of the surface electromyography signals obtained from the SENIAM electrodes during the dynamic tasks. | At study enrollment.
Fugl-Meyer Assessment score of the paretic lower limb. | At study enrollment.
  Maximum score is 34.
Passive ankle range of motion. | At study enrollment.
  This will be measured using a manual goniometer.

IPD SHARING:
Plan to Share IPD: No